CLINICAL TRIAL: NCT05763277
Title: Developing Atezolizumab-Bevacizumab Treatment Response Early Prediction Model in Advanced Hepatocellular Carcinoma Patients
Brief Title: Ate-Bev Early Response Prediction Model in Advanced HCC
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong-Hoon Lee, Professor, Seoul National University Hospital
Other Study IDs: 2206-066-1332
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Hepatocellular Carcinoma; Atezolizumab-bevacizumab; Response Evaluation
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ate-Bev: Individuals diagnosed with advanced hepatocellular carcinoma and treated with atezolizumab-bevacizumab between the ages of 18-80 were included. According to the recommendations of the American Society of Clinical Oncology-Friends of Cancer Research Organ Dysfunction, patients with comorbidities were excluded.
  Interventions: Diagnostic Test: Early response evaluation

INTERVENTIONS:
Diagnostic Test: Early response evaluation — Atezolizumab and bevacizumab are administered every three weeks, and before to the second treatment cycle, blood tests and imaging tests are conducted (week 5). This precedes the standard response evaluation (week 9-12).

SUMMARY:
The prognosis of hepatocellular carcinoma is poor compared to other carcinomas. Many drugs have recently been developed, and recently, atezolizumab-bevacizumab treatment was superior to sorafenib, the conventional treatment for advanced hepatocellular carcinoma. However, there is no information on the evaluation on the evaluation of treatment response for atezolizumab-bevacizumab combination therapy compared to atezolizumab alone or bevacizumab alone. Therefore, this study aimed to create a predictive model that can detect treatment response at an early stage.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed with advanced hepatocellular carcinoma and who were scheduled to receive atezolizumab-bevacizumab as the first-line therapy
* Patients willing to participate in this study

Exclusion Criteria:

* Individuals with a history of severe contrast allergy
* Individuals with severe comorbidities (according to the American Society of Clinical Oncology-Friends of Cancer Research Organ Dysfunction.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed with advanced hepatocellular carcinoma and who were scheduled to receive atezolizumab-bevacizumab as the first-line therapy in a single tertiary hospital are included.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2022-07-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
progression free survival | the follow up will be continued until June 22th 2025.
  the index date is the date of treatment with atezolizumab and bevacizumab, and the event is either death or tumor progression of the tumor.

SECONDARY OUTCOMES:
Overall survival | the follow up will be continued until June 22th 2025.
  the index date is the date of treatment with atezolizumab and bevacizumab, and the event is death.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea